CLINICAL TRIAL: NCT07361549
Title: Localized Injection of Lidocaine Via the Middle Meningeal Artery for Intractable Headache Treatment: A Randomized, Double-Blinded, Parallel Phase 2 Clinical Trial
Brief Title: Localized Injection of Lidocaine Via the Middle Meningeal Artery for Intractable Headache Treatment
Acronym: LIGHT 2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daniel A Tonetti, MD (Other)
Responsible Party: Sponsor-Investigator, Daniel A Tonetti, MD, Assistant Professor of Neurological Surgery, The Cooper Health System
Organization: The Cooper Health System (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-279
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Refractory Migraine; Headache
Keywords: headache; migraine; lidocaine; middle meningeal artery
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Lidocaine; Pharmaceutical Preparations; Sodium Chloride; Fluid Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Intra-arterial lidocaine
  Interventions: Drug: Lidocaine (drug)
- Sham (Sham Comparator): Intra-arterial saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine (drug) — Intra-arterial lidocaine infusion into bilateral middle meningeal arteries
  Other Names: Xylocaine
  Arms: Treatment
Drug: Saline — Intra-arterial saline infusion into bilateral middle meningeal arteries
  Other Names: Fluids
  Arms: Sham

SUMMARY:
The goal of this clinical trial is to test whether injecting lidocaine into two blood vessels of the brain can help treat chronic headaches (migraines)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Referred for diagnostic angiography
* Diagnosis of intractable migraine
* Written informed consent able to be obtained from subject

Exclusion Criteria:

* Baseline HIT-6 score less than 60 (severe)
* Pregnant, breastfeeding, or unwilling to practice contraception during participation in the study
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Concomitant intracranial pathology (eg, intracranial malignancy)
* Known hypersensitivity and/or contraindication to lidocaine or local anesthetics of the amide type
* Taking chronic medications that, when co-administered with lidocaine and other local anesthetics, are at increased risk of developing methemoglobinemia (nitrates/nitrites, local anesthetics, antineoplastic agents, antibiotics, antimalarials, anticonvulsants, acetaminophen, metoclopramide, quinine, sulfasalazine)
* Known contraindications for angiography (eg, ESRD not requiring hemodialysis). Patients with contrast allergy with be premeditated with diphenhydramine and steroids.
* Contraindication to anesthetic agents used for conscious sedation/monitored anesthesia care (MAC)
* Concurrent participation in another research protocol for investigation of an experimental therapy
* Per DSA imaging, presence of a cerebrovascular pathology known to cause headache (eg, arteriovenous malformation, dural arteriovenous fistula)
* Per DSA imaging, presence of anastomosis or anatomical variation (eg, branches of middle meningeal artery) that could lead to increased procedural risk
* Per DSA imaging, lack of endovascular access to either middle meningeal artery, or origin of the middle meningeal artery other than from the external carotid artery
* Known or suspected inability to adhere to study protocol or protocol requirements, as per discretion of the Investigator or treating provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Change in Headache Impact Test-6 Scores | From baseline to 4 week follow-up
  Difference in Headache Impact Test-6 Scores, with larger decreases in scores correlating with improvement in symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Koneru, MD, Study Chair — The Cooper Health System
Locations (1):
- Cooper University Health Care, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No